CLINICAL TRIAL: NCT01652066
Title: Effect of a Mixture of Probiotics ( Lactobacillus Gasseri PA16/8,Bifidobacterium Longum SP07/3, Bifidobacterium Bifidum MF 20/5) on the Antigen Specific Antibody Response in a Influenza Vaccination Model of Healthy Adult
Brief Title: Effect of a Mixture of Probiotics on the Antigen Specific Antibody Response in a Influenza Vaccination Model of Healthy Adults
Acronym: PROBIMMUNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Medication Familiale (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2011-A00225-36
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Enhancement of Protective Antibody Response After Probiotic Consumption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): oral consumption, once per day in the morning, fasting, with a glass of water
  Interventions: Dietary Supplement: Mixture of probitiocs
- Mixture of probiotics (Experimental): at least 10x7 cfu/tablet of a mixture of probiotics
  oral consumption, once per day in the morning, fasting, with a glass of water
  Interventions: Dietary Supplement: Mixture of probiotics

INTERVENTIONS:
Dietary Supplement: Mixture of probiotics — effect of the consumption a mixture of probiotics ( dietary supplement tablet - dosage at least 10x7 cfu/g) during 7 weeks , once a day , healthy volonteers ) on the antigen specific antibody respense
  Arms: Mixture of probiotics
Dietary Supplement: Mixture of probitiocs — effect of the consumption a mixture of probiotics ( dietary supplement tablet - dosage at least 10x7 cfu/g) during 7 weeks , once a day , healthy volonteers ) on the antigen specific antibody respense
  Arms: Placebo

SUMMARY:
the aim of the study is to get evidence for an enhancement of immune status in subjects after probiotics mixture consumption ( lactobacillus gasseri PA 16/8, Bifidobacterrium longum SP 07/3, Bifidobacterium bifidum MF 20/5) based on influenza vaccination model - compared to placebo.

DETAILED DESCRIPTION:
probiotics are "live microorganisms which when administered in adequate amounts confer a health benefit on the host" . many health effects are associated with probiotics , but various degrees of evidence support the benefits associated to probiotics consumption . Impact on defences and the immune system has been shown with several strains and this may result in improved protection against some infections or improvment of vaccine efficacy .

In its scientific requirments for health claims related to immune function, EFSA indicates that it is generally accepted that higher vaccination responses are beneficial.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female adult
* between 18 and 60 years old non menopausal female( with effective contraception)
* female non pregnant- not wishing to be pregnat during the study capable to respect the protocol
* affialted to the social security system aggreeing to be registered in the national fileof volunteers

Exclusion Criteria:

* food allergy( component of the experimental product- vaccines)
* manifestation of allergy
* vaccinated against flu during the 2 previous winters
* Food allergy, allergy to one of the component of the experimental products or allergy to one of the component of the flu vaccine;
* Subject displaying manifestation of allergy or being treated for these;
* Subject vaccinated against flu during the 2 previous winter (winter 2009-2010 and winter 2010-2011);
* Subject who had symptoms evocating flu during the previous winter (winter 2010-2011);
* Subject immunodepressed;
* Subject with immunomodulatory treatment;
* Subject who received a treatment resulting in systemic immunossuppression or local immunosuppression at pulmonary level, for at least 1 week during the last 3 months before inclusion (V1);
* Subject with auto-immune disease;
* Subject with inflammatory and chronic diseases;
* Subject with on-going antibiotics treatment at the time of the inclusion;
* Subject not agree to stop his/her usual probiotics supplementation during the study;
* Use of medication which could interfere with the study in the investigator's opinion (antibiotics, etc…);
* Any health condition for which the influenza vaccine is not recommended;
* Subject having received any other vaccine within one month prior to enrolment or intent to receive any other vaccination during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
geographic mean of the increase of antibody titreq against at least one flu strain among the 3 forming the flu vaccine ( H1N1, H3, N and B ) within 3 weeks after flu vaccination | inclusion-W 4-W 7

SECONDARY OUTCOMES:
seroprotection of the population of volunteers geometric mean of the increase of antibody titres seroprotection in the subset population non sero-protected at V1 | inclusion- W4- W7

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Nantes, France